CLINICAL TRIAL: NCT01010334
Title: Randomized Study of Patients (Patient Choice) Who Are Not Eligible for Variations of Standard of Care Protocols When Treated Either on Best Standard of Care Pathways or Per a Protocol Arm That They Failed to Enroll to
Brief Title: Comparison of Standard of Care or Treatment on Protocol
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI deparature and very low (<2%) accrual rate.(No results required)
Sponsor: New Mexico Cancer Research Alliance (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: INST 0813; NCI-2011-02680 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2009-07-24; First posted 2009-11-10 (Estimated); Last update posted 2013-08-14 (Estimated); Status verified 2013-08

CONDITIONS: Stomach Cancer; Esophageal Cancer; Bladder Cancer; Skin Cancer; Lung Cancer; Uterine Cancer; Ovarian Cancer
Keywords: INST 0813; Standard of Care
MeSH Terms: conditions — Stomach Neoplasms; Esophageal Neoplasms; Urinary Bladder Neoplasms; Skin Neoplasms; Lung Neoplasms; Uterine Neoplasms; Ovarian Neoplasms | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Active Comparator): Standard of Care Treatment
  Interventions: Other: standard of care
- Arm 2 (Experimental): Treatment Arm of a separate protocol (physician discretion)
  Interventions: Other: standard of care

INTERVENTIONS:
Other: standard of care — All patients failing to enroll in a specific therapeutic research protocol using FDA approved drugs or CTMS accepted therapies will be screened for this study. Patients will be randomized (Patient own choice) to either standard of care described in the NCCN guidelines and published as peer-reviewed phase II or III studies which show an efficacy, OR to one of the arms of the protocol they failed to enroll in, as determined by the treating physician.
  Other Names: Standard of Care therapy (disease site based); VARIIOUS experimental therapies (based on protocol for which pt failed eligibility)

SUMMARY:
Patient will choose to either receive the standard of care according to National Comprehensive Cancer Network (NCCN) or approved guidelines for their condition or to be treated according to one arm of the protocol that they could not be enrolled on. The selection of the arm will be at physician discretion.

DETAILED DESCRIPTION:
All patients failing to enroll in a specific therapeutic research protocol using FDA approved drugs or CTMS accepted therapies will be screened for this study. Patients will be randomized (Patient own choice) to either standard of care described in the NCCN guidelines and published as peer-reviewed phase II or III studies which show an efficacy or to one of the arms of the protocol they fail to enroll in, as determined by the treating physician.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a cancer requiring chemotherapy or radiotherapy

Exclusion Criteria:

* Inability to comply with study and/or follow-up procedures
* Any contraindication per the FDA notice to the selected drugs
* Pregnant (positive pregnancy test) or lactating. No effective means of contraception (men and women) in subjects of child-bearing potential

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2009-03; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Number of courses delivered (relative dose intensity for adjuvant studies) | 6 months

SECONDARY OUTCOMES:
Response rate | 6 months
Progression- or disease-free survival (for metastatic disease) | 6 months
Overall survival | 6 months
Describe all adverse events of grade > 3 and Serious Adverse Events | 6 months
Measure quality of life using a FACT G tool, before and at best response and at the end of the treatment | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Claire Verschraegen, MD, Principal Investigator — University of New Mexico Cancer Center
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States